CLINICAL TRIAL: NCT05564832
Title: Pharmacological Treatment of Presbyopia by Pilocarpine 1.25% Eye Drops
Brief Title: Pharmacological Treatment of Presbyopia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamideh Sabbaghi, Assistant Professor, Shahid Beheshti University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.SBMU.ORC.REC.1401.005
Record Dates: First submitted 2022-09-17; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Near Vision
MeSH Terms: conditions — Myopia | interventions — Pilocarpine; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilocarpine Therapy (Experimental): The right eyes of 45 patients will be treated by Biocarpine® and Vuity® eye drops. They will be considered as the case group,
  Interventions: Drug: Pilocarpine 1.25% Eye drop
- Without Pilocarpine Therapy (No Intervention): The left eyes of the patients will be defined as the controls.

INTERVENTIONS:
Drug: Pilocarpine 1.25% Eye drop — One millimeter of pilocarpine eye drop (Bakhtarbiochemistry Company, Iran) contains pilocarpine hydrochloride 1.25% (12.5 mg) as an active ingredient, equivalent to 1.06% (10.6 mg) pilocarpine free-base. The medication preservative is 0.0075% benzalkonium chloride. Inactive ingredients in the ophthalmic are boric acid, sodium citrate dihydrate, sodium chloride, purified water. Another pilocarpine eye drop was Vuity® (1.25% pilocarpine; Allergan company) contains the active intergradients of pilocarpine hydrochloride 1.25% (12.5 mg/mL), equivalent to 1.06% (10.6 mg/mL) pilocarpine free-base and the preservative agents was 0.0075% benzalkonium chloride.
  Arms: Pilocarpine Therapy

SUMMARY:
In this clinical trial, a total of 75 presbyopic patients in the age range of 40 to 60 years old will be participated. The right eyes of 45 patients will be treated by Biocarpine® and they will be considered as the case group, their left eyes will be defined as the controls. In another case group, the right eyes of 30 patients will received Vuity® eye drops and their left eyes will be considered as controls.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with the best corrected visual acuity (BCVA) better than 0.3LogMAR
* Patients with the symptom of blurred vision at near distance

Exclusion Criteria:

Patients with amblyopia, cataract, corneal opacity, glaucoma, intraocular surgery, eye troma, congenital pupil anomalies and those with the history of headache and allergy to the eye drop will be excluded from the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
The changes of near vision after one hour following pilocarpine eye drop | baseline to one hour after pilocarpine insillation
  The near vision will be measured based on the LogMAR vision at a distance of 33cm before and one hour after instillation of 1.25% pilocarpine eye drop.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamideh Sabbaghi, Tehran, Iran